CLINICAL TRIAL: NCT01708356
Title: Cycling, Air Pollution and Health
Acronym: CAPaH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H10-00902; H1008-111481/001/XSB (Other: UBC CREB)
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Endothelial Dysfunction; Endothelial Function; Cardiovascular Physiological Phenomena
Keywords: Air Pollution; Particulate Matter; Exercise; Respiratory Rate; Inflammation; Oxidative Stress; Plethysmography
MeSH Terms: conditions — Motor Activity; Inflammation

ARMS (1):
- Normal cycling (Experimental): Cycling on a residential and downtown route (crossover design)
  Interventions: Behavioral: Cycling on a residential route

INTERVENTIONS:
Behavioral: Cycling on a residential route

SUMMARY:
Introduction: Cycling is currently promoted at the municipal, provincial and national level as a form of active transportation that increases physical activity while at the same time reducing traffic congestion, traffic-related air pollution and greenhouse gas emissions. While at a population level the health benefits of exercise via cycling are estimated to substantially exceed any health impacts related to air pollution exposure and injuries from traffic accidents , cyclists are known to experience elevated exposures to traffic-related air pollutants. Combined with exposure to elevated concentrations of air pollutants, cyclists also are subject to substantially increased inhaled doses due to their level of exertion and consequently increased inhalation rate. Therefore, given that cyclists experience exposures to relatively high concentrations of traffic-related air pollutants and that their inhalation of these pollutants is increased, it is important to evaluate the potential health impacts of this scenario. Research on the potential health impacts related to exercise (cycling) and urban air pollution exposure can help inform public communication strategies related to air quality and its health impacts. In addition, as our previous work suggests substantial variability in air pollution exposures to cyclists that is related to the route type and the levels of traffic along cycling routes, there is potential for transportation planners to promote increased cycling by enhancing infrastructure while at the same time developing routes that also minimize exposure to air pollution. The cyclist population is also interested in information regarding the air pollution exposures and potential health impacts related to cycling.

The objective of this study is to investigate the relationship between traffic-related air pollution exposure, and respiratory and cardiovascular health impacts in commuting cyclists. Specifically, the investigators propose to:

1. determine commuting cyclists' exposure to traffic-related air pollutants (PM 2.5, PM10, ultrafine particulate, black carbon) while cycling along two different bicycle routes in the city of Vancouver;
2. estimate the pollutant dose received by each cyclist, and relate this to the health effects observed; and
3. determine if there is a change in lung function, endothelial function, and C-reactive protein level related to the level of air pollution exposure and dose

ELIGIBILITY:
Inclusion Criteria:

* Age 19- 39
* male or female
* able to bicycle comfortably on city streets for 1 hour

Exclusion Criteria:

* Smokers of any substance (smoking more than 1x every 2 weeks)
* Must be of height to safely ride a test bike (<5'2", >6'5" )
* Diagnosed asthma or active allergy (hav fever) symptoms
* Irregular menstrual cycle, pregnant, breastfeeding, non-monocyclic contraceptive medication or device
* Taking medication for heart or lung condition
* Answers yes to any questions on physical activity readiness questionnaire (PAR-Q)
* requires pain medication daily
* visual or hearing impairment that prevents safe cycling on streets with motor vehicles

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function, as measured by peripheral arterial tonometry (EndoPAT) score of reactive hyperemia index (RHI) | Baseline (1 hour pre-expousre) and 1 hour post- exposure (plus or minus 30 minutes) to a bicycle ride in an urban environment outdoors

SECONDARY OUTCOMES:
Change in lung function (using spirometry to assess lung function values) | Baseline (1 hour pre-exposure) and 1 hour post- exposure (plus or minus 30 minutes) to a bicycle ride in an urban environment outdoors

OTHER OUTCOMES:
Change in blood levels of C-reactive protein (a marker of systemic inflammation) | Baseline (1 hour pre-exposure) and 1 hour post- exposure (plus or minus 30 minutes) to a bicycle ride in an urban environment outdoors
Change in blood levels of Interleukin-6 (a marker of systemic inflammation) | Baseline (1 hour pre-exposure) and 1 hour post- exposure (plus or minus 30 minutes) to a bicycle ride in an urban environment outdoors
Change in blood levels of 8-hydroxy-2'-deoxyguanosine (8-OHdG)(a marker of oxidative stress) | Baseline (1 hour pre-exposure) and 1 hour post- exposure (plus or minus 30 minutes) to a bicycle ride in an urban environment outdoors

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brauer, ScD, Principal Investigator — The University of British Columbia
Locations (1):
- Air Pollution Exposure Lab, Vancouver General Hospital through the School of Population and Public Health, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Cole CA, Carlsten C, Koehle M, Brauer M. Particulate matter exposure and health impacts of urban cyclists: a randomized crossover study. Environ Health. 2018 Nov 14;17(1):78. doi: 10.1186/s12940-018-0424-8. PMID 30428890